CLINICAL TRIAL: NCT07234903
Title: ARC-IM Therapy To Support and Promote Recovery of Ambulatory Functions in People With Subacute and Chronic Spinal Cord Injury
Acronym: EIGER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Principal Investigator, Jocelyne Bloch, Professor, Centre Hospitalier Universitaire Vaudois
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EIGER
Record Dates: First submitted 2025-09-01; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injury; SCI; SCI - Spinal Cord Injury; Subacute Spinal Cord Injury; Chronic Spinal Cord Injury; Spinal Cord Injury (SCI)
Keywords: SCI; Spinal Cord Injury; Epidural Electrical Stimulation; Spinal Cord Stimulation; ARC-IM Therapy
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Multicentric, two-arms, non-blinded, non-randomized, interventional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subacute SCI (Experimental): Participants having sustained the injury less than 6 weeks prior to baseline (subacute).
  Participants will be provided with the ARC-IM Therapy.
  Interventions: Device: ARC-IM Therapy
- Chronic SCI (Experimental): Participants having sustained the injury more than 1 year prior to enrollment (chronic).
  Participants will be provided with the ARC-IM Therapy.
  Interventions: Device: ARC-IM Therapy

INTERVENTIONS:
Device: ARC-IM Therapy — All participants will be treated with ARC-IM Therapy. The ARC-IM Lumbar System is intended to deliver electrical impulses to the lumbosacral region of the spinal cord to support ambulatory functions in people with SCI.

SUMMARY:
The EIGER study aims to evaluate the safety and preliminary efficacy of ARC-IM Therapy (Epidural Electrical Stimulation) to support and promote recovery of ambulatory functions, such as walking, in people with subacute and chronic spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

1. Must be at least 18 years old and no older than 65 years old at the time of enrollment.
2. Must be graded A, B, C, or D in the ASIA Impairment Scale (AIS).
3. Must have a SCI level at T10 or higher as determined by ISNCSCI, with the region extending 6 cm above the tip of the conus remaining anatomically intact as determined by MRI.
4. Must have sustained their injury either less than 6 weeks prior to baseline (Group "Subacute SCI"), or more than 1 year prior to enrollment (Group "Chronic SCI").
5. Must be suffering from a SCI due to trauma.
6. Must have a stable medical, physical and psychological condition as considered by the investigators and the delegated specialists.
7. Must have residual upper limb function to use the arms for weight bearing support (as determined by functional demonstration).
8. Must be able to understand and interact with the study team in German, French or English.
9. Must agree to comply in good faith with all conditions of the study and to attend all scheduled appointments.
10. Must provide Informed Consent as documented by signature prior to any study-related procedures.
11. Must have an acceptable or highly effective method of contraception for women of childbearing capacity.

Exclusion Criteria:

1. Must not be pregnant nor breastfeeding.
2. Must not have brain damage.
3. Must not have a history of epilepsy
4. Must not have participated in another clinical study using drugs or medical devices within the 30 days preceding and during the present study.
5. Must not have previously been injected with stem cells in the spinal cord.
6. Must not have any diseases and conditions that would increase the morbidity and mortality of SCI surgery.
7. Must not require ventilator support.
8. Must not have any existing contraindication to mobility functions (e.g., unhealed bone fractures, central nervous system disorder, peripheral nerve disorder, etc.).
9. Must not suffer from SCI from other etiology than trauma (ischemic, tumoral, autoimmune, etc.).
10. Must not have any anatomical limitations in the implantation area as judged by the investigators (e.g., spinal stenosis, limiting protrusions, post-traumatic bone damage at area of implantation).
11. Must not require the use of an intrathecal baclofen pump.
12. Must not have any active implanted devices.
13. Must not have any other conditions that would make the subject unable to participate in testing in the judgment of the investigators (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.).
14. Must not be the investigator him/herself, his/her family members, employees or other dependent persons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2032-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Serious Adverse Events and Adverse Events that are deemed related or possibly related to the study procedure or to ARC-IM Therapy, from implantation up to the end of the study. | Continuously throughout the study (up to 6 years)
  Assess the preliminary safety of ARC-IM Therapy in participants with subacute and chronic SCI.

SECONDARY OUTCOMES:
American Spinal Injury Association (ASIA) International Standards for the Neurological Classification of Spinal Cord Injury (ISNCSCI) | At Eligibility, and at 6 weeks, 16 weeks, 42 weeks post-surgery
  The ASIA ISNCSCI is a clinical examination used to assess the motor and sensory impairment and severity of a spinal cord injury.
10-Meter Walk Test (10MWT) | At Baseline, and at 6 weeks, 16 weeks, ad 42 weeks post-surgery
  The 10MWT assesses walking speed in meters per second over a short duration. It measures the time taken by the subjects to walk 10 meters. The test will be performed twice, at self-selected and at maximum velocity. Participants can use their habitual assistive device. The test will be conducted both with and without stimulation.
6-Minute Walk Test (6MWT) | At Baseline, and at 6 weeks, 16 weeks, and 42 weeks post-surgery
  The 6MWT assesses endurance by measuring the distance in meters a participant walks in 6 minutes. Participants can use their habitual assistive device and can take as many standing breaks as they need, but the timer will not be paused. This test will be conducted both with and without stimulation.
Timed Up and Go (TUG) | At Baseline, and at 6 weeks, 16 weeks, and 42 weeks post-surgery
  The TUG evaluates functional mobility. Participants begin seated, then stand up, walk 3 meters, turn around, walk back, and sit down. The time taken to complete the sequence is recorded. Assistive devices may be used if necessary. The test will be conducted both with and without stimulation.
Walking Index for Spinal Cord Injury version II (WISCI II) | At Baseline, and at 6 weeks, 16 weeks, and 42 weeks post-surgery
  The WISCI II assesses the extent and nature of assistance a person with SCI requires to walk, using an ordinal scale of 20 levels, ranging from the most severe impairment (level 0) to the least severe impairment (level 20). The level is determined based on the use of assistive devices, braces, and the physical assistance of one or more persons. The test will be conducted both with and without stimulation.
Spinal Cord Injury Functional Ambulation Inventory (SCI-FAI) | At Baseline, and at 6 weeks, 16 weeks, and 42 weeks post-surgery
  The SCI-FAI assesses functional walking ability. It is an observational gait assessment that includes 3 key domains of walking function, where 0 is the minimum and worst outcome: gait parameters (maximum score of 20 points), assistive device (each limb scored individually - maximum score of 14 points), and temporal distance (maximum score of 5 points). The test will be conducted both with and without stimulation.
Gait Analysis | At Baseline, and at 6 weeks, 16 weeks, and 42 weeks post-surgery
  Multifactorial gait analysis that relies on high-precision recordings of whole-body kinematics and kinetics of each gait cycle will be performed. The test will be conducted both with and without stimulation.
Goal Attainment Scale (GAS) | At Baseline, and at 6 weeks, 16 weeks, and 42 weeks post-surgery
  The GAS is used to evaluate the participant's progress toward one or more personalized goal(s), which are individually defined by the participant. Each goal is scored on a standardized scale ranging from -2 (outcome is much less than expected) to +2 (outcome is much more than expected), allowing to assess to which extent the goal is met. The form will be completed for both with and without stimulation condition.
Berg Balance Scale (BBS) | At Baseline, and at 6 weeks, 16 weeks, 42 weeks post-surgery
  The BBS assesses static and dynamic balance through 14 tasks, such as standing, reaching, and turning. Each item is scored on a 5-point scale (0-4) with higher scores meaning better ability to perform the assessed activity. Item scores are then summed, with a maximum score of 56. The use of assistive devices is not allowed. The test will be conducted both with and without stimulation.

OTHER OUTCOMES:
ARC-IM stimulation usage log | At 6 weeks, 16 weeks, 42 weeks post-surgery, and at the end of the study
  Independent use of the ARC-IM Lumbar System by study participants will be evaluated through analysis of the ARC-IM stimulation usage log.
Integration of ARC-IM Therapy within the standard-of-care | At 6 weeks, 16 weeks, and 42 weeks post-surgery
  Integration of ARC-IM Therapy within the standard-of-care for subacute SCI will be evaluated by quantifying its use within standard clinical mobility rehabilitation procedures. This will be achieved by extracting and comparing data of the Stimulation Usage Log and Participant's Calendar Log.
EES Evoked Muscle Response | Every 2 days during the mapping phase, and at 6 weeks, 16 weeks, and 42 weeks post-surgery
  Effect of ARC-IM Therapy on the modulation of the spinal cord will be evaluated through electrophysiological assessments that will quantify the muscle responses to EES and adaptation of these responses over time.
Function In Sitting Test for Spinal Cord Injury (FIST-SCI) | At Baseline, and at 6 weeks, 16 weeks, and 42 weeks after surgery
  Effect of ARC-IM Therapy on trunk stability will be evaluated using the FIST-SCI. The FIST-SCI assesses sitting balance. It evaluates sensory, motor, proactive, reactive, and steady state balance factors based on 14 items, each scored on an ordinal scale from 0 to 4, where 0 means complete assistance is needed to perform the task successfully, and 4 means can complete the task independently and successfully. The test will be conducted both with and without stimulation.
Modified Ashworth Scale (MAS) | At Baseline, and at 6 weeks, 16 weeks, and 42 weeks post-surgery
  Effect of ARC-IM Therapy on muscle tone will be evaluated using the MAS. The MAS assesses spasticity in a participant's upper and lower limb, by rating the resistance of a muscle to passive movement at a single joint on a 6-point nominal scale, where 0 means no increase in tone, and 5 means affected parts are rigid in flexion or extension. The clinical examination will be performed both with and without stimulation on different days at similar times. Antispastic medication and time points of test/medication intake will be documented.
Spinal Cord Assessment Tool for Spastic Reflexes (SCATS) | At Baseline, and at 6 weeks, 16 weeks, and 42 weeks post-surgery
  Effect of ARC-IM Therapy on muscle tone will be evaluated using the SCATS. The SCATS assesses 3 types of spastic motor behaviors in SCI patients - clonus, flexor spasms, and extensor spasms. The clinical examination will be performed both with and without stimulation. Antispastic medication and start time of the test will be documented for inter-test reliability.
Spinal Cord Injury - Quality of Life Short form (SCI-QoL SF) | At Baseline, and at 6 weeks, 16 weeks, and 42 weeks post-surgery
  Effect of ARC-IM Therapy on quality of life will be evaluated with the SCI-QoL SF. The SCI-QoL SF is a PROM for individuals with SCI. It is divided into 4 domains (emotional health, physical-medical health, social participation, physical functioning) with a selection of 22 subdomains. Each subdomain has several items. The participant rates each item with a number between 1 and 5 according to the extent to which the statement it contains applies to them. Each subdomain is scored separately. The higher the score, the higher the participant's perceived quality of life.
EuroQol 5-Dimension 5-Level questionnaire (EQ-5D-5L) | At Baseline, at 6 weeks, 16 weeks, and 42 weeks post-surgery, and yearly until the end of study
  Effect of ARC-IM Therapy on quality of life for chronic SCI participants will be evaluated with the EQ-5D-5L questionnaire. The EQ-5D-5L is a PROM that describes the patient's health state for five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Patient Global Impression of Change (PGI-C) | At 6 weeks, 16 weeks, and 42 weeks post-surgery
  Effect of ARC-IM Therapy on the subjective change of overall status will be evaluated with the PGI-C. The PGI-C is a single-item questionnaire to measure the change of clinical status, injury severity, or injury improvement, and evaluate the response of a condition to the given therapy. It is a 7-point scale where the participant rates his/her improvement or deterioration on a scale from "1 = very much improved" to "7 = very much worse".
Spinal Cord Independence Measure (SCIM) III | At Baseline, and at 6 weeks, 16 weeks, and 42 weeks post-surgery
  Effect of ARC-IM Therapy on functional independence in daily living will be evaluated with the SCIM III score. The SCIM III is a disability score that addresses functional ability in daily living in people with SCI. Three specific areas are assessed: self-care (0-20 points), respiration and sphincter management (0-40 points), and mobility (0-40 points). The form will be filled out as per stimulation use of the participant in his/her daily life activities for with or without stimulation condition. Total score ranges between 0 and 100 points, with higher scores reflecting greater independence.
System Usability Scale (SUS) | At 6 weeks, 16 weeks, and 42 weeks post-surgery
  The SUS is a standardized post-usability test questionnaire comprised of 10 Likert-scale questions used to evaluate the usability of the investigational system. To collect the SUS score, participants rate how strongly they agree or disagree with statements on a 1 (strongly disagree) to 5 (strongly agree) scale.
EMSCI Pain Assessment Form (EPAF) | At Baseline, and at 6 weeks, 16 weeks, and 42 weeks post-surgery
  Effect of ARC-IM Therapy on pain will be evaluated with the EPAF. The EPAF is used for classification of existing pain problems in people with SCI. The clinical assessment form consists of 12 items and follows the international guidelines and recommendations for the clinical documentation and assessment of pain in SCI. One overall form will be completed summarizing with and without stimulation condition.
Dual-Energy X-Ray Absorptiometry (DEXA) | At Baseline and at 42 weeks post-surgery
  Effect of ARC-IM Therapy on bone mineral density will be evaluated using DEXA. Participants will lie in a supine position during the scan, following standardized protocols.
Quantitative Computed Tomography (QCT)-Scan | At Eligibility and at 42 weeks post-surgery
  Effect of ARC-IM Therapy on muscle mass will be evaluated using QCT-Scan. The QCT-Scan is used to assess muscle mass by providing high-resolution cross-sectional images of the thigh and the trunk. It allows for precise measurement of muscle volume and composition. Participants will undergo the scan in a supine position, and standardized protocols will be used to ensure consistency across time points.
Additional User Feedback | At 6 weeks, 16 weeks, and 42 weeks post-surgery
  The Additional User Feedback is a form designed to collect qualitative feedback from participants regarding their interaction with the ARCIM Lumbar System. It includes rating items to evaluate satisfaction (from "not satisfied at all" to "very satisfied") and open-ended questions addressing ease of use, satisfaction with system components such as battery life, charging time, connection stability, and overall comfort during use.

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyne Bloch, Prof. Dr. MD, Principal Investigator — CHUV; Björn Zörner, PD Dr. med. Dr. sc. nat., Principal Investigator — SPZ
Locations (2):
- Switzerland (2):
  - Schweizer Paraplegiker-Zentrum (SPZ), Nottwil, Canton of Lucerne
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud

REFERENCES:
- [Background] Capogrosso M, Wenger N, Raspopovic S, Musienko P, Beauparlant J, Bassi Luciani L, Courtine G, Micera S. A computational model for epidural electrical stimulation of spinal sensorimotor circuits. J Neurosci. 2013 Dec 4;33(49):19326-40. doi: 10.1523/JNEUROSCI.1688-13.2013. PMID 24305828
- [Background] Kathe C, Skinnider MA, Hutson TH, Regazzi N, Gautier M, Demesmaeker R, Komi S, Ceto S, James ND, Cho N, Baud L, Galan K, Matson KJE, Rowald A, Kim K, Wang R, Minassian K, Prior JO, Asboth L, Barraud Q, Lacour SP, Levine AJ, Wagner F, Bloch J, Squair JW, Courtine G. The neurons that restore walking after paralysis. Nature. 2022 Nov;611(7936):540-547. doi: 10.1038/s41586-022-05385-7. Epub 2022 Nov 9. PMID 36352232
- [Background] Wagner FB, Mignardot JB, Le Goff-Mignardot CG, Demesmaeker R, Komi S, Capogrosso M, Rowald A, Seanez I, Caban M, Pirondini E, Vat M, McCracken LA, Heimgartner R, Fodor I, Watrin A, Seguin P, Paoles E, Van Den Keybus K, Eberle G, Schurch B, Pralong E, Becce F, Prior J, Buse N, Buschman R, Neufeld E, Kuster N, Carda S, von Zitzewitz J, Delattre V, Denison T, Lambert H, Minassian K, Bloch J, Courtine G. Targeted neurotechnology restores walking in humans with spinal cord injury. Nature. 2018 Nov;563(7729):65-71. doi: 10.1038/s41586-018-0649-2. Epub 2018 Oct 31. PMID 30382197
- [Background] Rowald A, Komi S, Demesmaeker R, Baaklini E, Hernandez-Charpak SD, Paoles E, Montanaro H, Cassara A, Becce F, Lloyd B, Newton T, Ravier J, Kinany N, D'Ercole M, Paley A, Hankov N, Varescon C, McCracken L, Vat M, Caban M, Watrin A, Jacquet C, Bole-Feysot L, Harte C, Lorach H, Galvez A, Tschopp M, Herrmann N, Wacker M, Geernaert L, Fodor I, Radevich V, Van Den Keybus K, Eberle G, Pralong E, Roulet M, Ledoux JB, Fornari E, Mandija S, Mattera L, Martuzzi R, Nazarian B, Benkler S, Callegari S, Greiner N, Fuhrer B, Froeling M, Buse N, Denison T, Buschman R, Wende C, Ganty D, Bakker J, Delattre V, Lambert H, Minassian K, van den Berg CAT, Kavounoudias A, Micera S, Van De Ville D, Barraud Q, Kurt E, Kuster N, Neufeld E, Capogrosso M, Asboth L, Wagner FB, Bloch J, Courtine G. Activity-dependent spinal cord neuromodulation rapidly restores trunk and leg motor functions after complete paralysis. Nat Med. 2022 Feb;28(2):260-271. doi: 10.1038/s41591-021-01663-5. Epub 2022 Feb 7. PMID 35132264